CLINICAL TRIAL: NCT04965870
Title: A Retrospective Observational Study of Trifluridine/ Tipiracil (TAS-102) in Chemorefractory Metastatic Colorectal Cancer (mCRC) in Greece. Real World Data on Clinical Benefit.
Brief Title: A Study of Trifluridine/ Tipiracil in Chemorefractory mCRC in Greece
Acronym: RETRO-TAS
Status: Completed | Type: Observational
Sponsor: Hellenic Study Group of Psychoneuroimmunology in Cancer (Network)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-01
Record Dates: First submitted 2021-06-28; First posted 2021-07-16 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Trifluridine/Tipiracil — Trifluridine/ Tipiracil is an oral combination of an antineoplastic thymidine-based nucleoside analogue, trifluridine, and the thymidine phosphorylase (TPase) inhibitor, tipiracil hydrochloride.
  Other Names: FTD/TPI; TAS 102

SUMMARY:
Collection of real world data on the clinical efficacy of trifluridine/ tipiracil (FTD/TPI) in the Greek population.

DETAILED DESCRIPTION:
The aim of this analysis is to record clinical practice and to collect real world data on the clinical efficacy of trifluridine/ tipiracil (FTD/TPI) in the Greek population. Main objectives include to assess physician's choice of treatment in chemoresistant metastatic colorectal cancer with FTD/TPI in third line and beyond In addition, the clinicopathologic features related to metastatic colorectal cancer (focus on molecular profile), duration of treatment, dose modification and toxicity will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically confirmed metastatic colorectal cancer
* Available data on previous chemotherapy lines

Exclusion Criteria:

No exclusion criteria have been established for this observational and retrospective study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Greek patients with mCRC
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Retrospective data analysis from January 2018 to at least 3 months prior to being included in the study.
  PFS is defined as the time interval from initiation of treatment to the first date of documented tumor progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival | Retrospective data analysis from January 2018 to at least 3 months prior to being included in the study.
  Overall survival is defined as the time interval from initiation of treatment to the date of death due to any cause.
Progression Free Survival rate at 6 and 8 months | Retrospective data analysis from January 2018 to at least 3 months prior to being included in the study.
  PFS rate at 6 and 8 months corresponding to the percentage of patients surviving without any documented progression of the disease at 6 and 8 months after treatment initiation.
Disease Control Rate | Retrospective data analysis from January 2018 to at least 3 months prior to being included in the study.
  The DCR is defined as the proportion of patients with objective evidence of complete response (CR), the proportion of patients with objective evidence of partial response (PR), and the proportion of patients with objective evidence of stable disease (SD).

CONTACTS AND LOCATIONS:
Overall Officials: ANNA KOUMARIANOU, PhD, Principal Investigator — 4th Department of Internal Medicine, Attikon University Hospital
Locations (8):
- Greece (8):
  - University General Hospital of Heraklion (PAGNI), Heraklion, Crete
  - General Hospital "Venizeleio - Pananio", Heraklion, Crete
  - Athens Medical Group, Athens
  - General Oncological Hospital "Agioi Anargyroi", Athens
  - Agios Savvas Cancer Hospital, Athens
  - Attikon University Hospital, Athens
  - Anticancer Hospital "METAXA", Piraeus
  - Bioclinic, Thessaloniki

IPD SHARING:
Plan to Share IPD: No